CLINICAL TRIAL: NCT01245270
Title: A Single Supplement of a Standardised Bilberry Extract (36% (w/w) Anthocyanins) Modifies Glycaemic Response in Persons With Type 2 Diabetes Controlled by Diet and Lifestyle.
Brief Title: A Single Supplement of a Standardised Bilberry Extract Modifies Glycaemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REC 10/S0801/54; 902 (Other: Rowett institute code)
Record Dates: First submitted 2010-11-16; First posted 2010-11-22 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
Keywords: anthocyanin; blaeberries; bilberries; blueberries; mirtoselect; glucose AUC
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vaccinium myrtillus extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilberry capsule first, then control cap (Experimental): Volunteers will be given a single capsule of 0.47 grams of mirtoselect (a concentrated bilberry extract) followed by a 14 day washout period then a single control placebo capsule.
  First Intervention (1 day), Washout (14 days), Second Intervention (1 day)
  Interventions: Dietary Supplement: Bilberry capsule first, then control cap
- Control capsule first, then bilberry cap (Experimental): Volunteers will be given a single control placebo capsule followed by a 14 day washout period the a single capsule of 0.47 grams of mirtoselect (a concentrated bilberry extract)
  First Intervention (1 day), Washout (14 days), Second Intervention (1 day)
  Interventions: Dietary Supplement: Control capsule first then bilberry cap

INTERVENTIONS:
Dietary Supplement: Bilberry capsule first, then control cap — Male subjects aged >40 and <70 years, with type 2 diabetes controlling their diabetes by diet alone closely matched for adiposity as determined by waist circumference (n=8).
  Volunteers will be randomised double blinded into two groups (n=4 per group) and given a single capsule of either 0.47 grams of a bilberry extract (mirtoselect provided by Indena S.p.A (http://www.mirtoselect.info/) or a control capsule. Following a two week wash out period the volunteers will be asked to take a second single capsule of either of 0.47 grams of mirtoselect or a control capsule in a cross over study, the opposite of what they took the first time.
  Arms: Bilberry capsule first, then control cap
Dietary Supplement: Control capsule first then bilberry cap — Male subjects aged >40 and <70 years, with type 2 diabetes controlling their diabetes by diet alone closely matched for adiposity as determined by waist circumference (n=8).
  Volunteers will be randomised double blinded into two groups (n=4 per group) and given a single capsule of either 0.47 grams of a bilberry extract (mirtoselect provided by Indena S.p.A (http://www.mirtoselect.info/) or a control capsule. Following a two week wash out period the volunteers will be asked to take a second single capsule of either of 0.47 grams of mirtoselect or a control capsule in a cross over study, the opposite of what they took the first time.
  Arms: Control capsule first, then bilberry cap

SUMMARY:
Dietary strategies for alleviating health complications associated with type 2 diabetes (T2D) are being pursued as alternatives to pharmaceutical interventions. Berries such as bilberries that are rich in polyphenols may influence carbohydrate digestion and absorption and thus postprandial glycaemia. In addition berries have been reported to alter incretins as well as to have anti-oxidant and anti-inflammatory properties that may also affect postprandial glycaemia. This study investigated the acute affect of a standardised bilberry extract on glucose metabolism in T2D.

Eight male volunteers with T2D controlling their diabetes by diet and lifestyle alone were given a single oral capsule of either 0.47g standardized bilberry extract (36% (w/w) anthocyanins) which equates to ∼50 g of fresh bilberries or placebo followed by a polysaccharide drink (equivalent to 75 g glucose) in a double blinded cross over intervention with a two week washout period.

This study demonstrates that the ingestion of a concentrated bilberry extract reduces postprandial glycaemia and insulin in volunteers with T2D. The most likely mechanism for the lower glycaemic response involves reduced rates of carbohydrate digestion and/or absorption.

DETAILED DESCRIPTION:
Dietary strategies for alleviating health complications, such as premature vascular disease, associated with type 2 diabetes (T2D) and obesity are actively being pursued as alternatives to pharmaceutical interventions. The genus Vaccinium (e.g. blueberry, bilberry, cranberry) has been used traditionally as a source of folk remedies for established diabetic symptoms.

Berries from this genus are enriched in anthocyanins, polyphenols recognized for their ability to provide and activate cellular antioxidant protection and inhibit inflammatory gene expression, activities that may contribute to the efficacy of the Vaccinium genus as ameliorators for type 2 diabetes. Consumption of a freeze-dried blueberry beverage for an 8 week period for example decreased plasma concentrations of the cardiovascular risk factors oxidized LDL, malondialdehyde and hydroxynonenal. In another trial, bioactives from blueberries improved insulin sensitivity in obese insulin-resistant men and women. In both these studies the investigators reported no change in inflammatory markers following supplementation although bilberry juice was shown to modulate plasma markers of inflammation C-reactive protein and IL-6 in subjects with increased risk of cardiovascular disease. These beneficial responses from human studies are supported by data that demonstrate long-term beneficial effects of anthocyanins from mouse models of obesity and diabetes.

There are also a number of studies in vitro and in vivo that suggest that polyphenols influence carbohydrate digestion and absorption, resulting in improved postprandial glycaemia in the short term. Polyphenols inhibit intestinal alpha glucosidase activity and glucose transport in vitro. In association with this, polyphenols administered to rodents suppress the elevation of blood glucose concentration after oral administration of mono- and di-saccharides. In humans, several studies have examined the effect of polyphenols on the post-prandial glycaemic response. In one study a test meal of mixed berry purée with sucrose showed a lower plasma glucose concentration after 15-30 min compared with a control matched for sugars.

Overall, evidence suggests that consuming edible berries, particularly from the genus Vaccinium, that have high concentrations of anthocyanins could provide a supplementary intervention to improve glycaemia in subjects with T2D or impaired glucose tolerance. The object of this study was to investigate whether a single supplementation with a standardised (36% w/w anthocyanins) concentrated bilberry extract could alter glucose metabolism in overweight/obese volunteers with impaired glucose intolerance or T2D compared with a control capsule matched for sugars and to explore the possible mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Aged >40 and <70
* Clinical diagnosis of Type 2 diabetes controlling their diabetes by diet alone
* All subjects must live in the Aberdeenshire area of Scotland

Exclusion Criteria:

* Medical exclusion criteria
* Clinical diagnosis of thromboembolic or coagulation disease
* Clinical diagnosis of unregulated thyroid disease
* Clinical diagnosis of kidney disease
* Clinical diagnosis of severe gastrointestinal disorders
* History of Alcohol or any other substance abuse

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hoggard, PhD, Principal Investigator — University of Aberdeen Rowett Institute of Nutrition and Health
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martineau LC, Couture A, Spoor D, Benhaddou-Andaloussi A, Harris C, Meddah B, Leduc C, Burt A, Vuong T, Mai Le P, Prentki M, Bennett SA, Arnason JT, Haddad PS. Anti-diabetic properties of the Canadian lowbush blueberry Vaccinium angustifolium Ait. Phytomedicine. 2006 Nov;13(9-10):612-23. doi: 10.1016/j.phymed.2006.08.005. Epub 2006 Sep 18. PMID 16979328
- [Background] Zafra-Stone S, Yasmin T, Bagchi M, Chatterjee A, Vinson JA, Bagchi D. Berry anthocyanins as novel antioxidants in human health and disease prevention. Mol Nutr Food Res. 2007 Jun;51(6):675-83. doi: 10.1002/mnfr.200700002. PMID 17533652
- [Background] Lau FC, Bielinski DF, Joseph JA. Inhibitory effects of blueberry extract on the production of inflammatory mediators in lipopolysaccharide-activated BV2 microglia. J Neurosci Res. 2007 Apr;85(5):1010-7. doi: 10.1002/jnr.21205. PMID 17265471
- [Background] DeFuria J, Bennett G, Strissel KJ, Perfield JW 2nd, Milbury PE, Greenberg AS, Obin MS. Dietary blueberry attenuates whole-body insulin resistance in high fat-fed mice by reducing adipocyte death and its inflammatory sequelae. J Nutr. 2009 Aug;139(8):1510-6. doi: 10.3945/jn.109.105155. Epub 2009 Jun 10. PMID 19515743
- [Result] Hoggard N, Cruickshank M, Moar KM, Bestwick C, Holst JJ, Russell W, Horgan G. A single supplement of a standardised bilberry (Vaccinium myrtillus L.) extract (36 % wet weight anthocyanins) modifies glycaemic response in individuals with type 2 diabetes controlled by diet and lifestyle. J Nutr Sci. 2013 Jul 24;2:e22. doi: 10.1017/jns.2013.16. eCollection 2013. PMID 25191571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight male volunteer subjects with T2D controlled by diet and lifestyle alone or with impaired glucose tolerance were recruited from the Aberdeen area of the UK. Subjects were only included if they were not on any special religious or prescribed diet and had a stable weight.
Groups:
- Single Control Capsule First Then Bilberry Capsule; Single Bilberry Capsule First Then Control Capsule: In a cross-over design, volunteers (n 8) were randomised and double-blinded into two groups matched for BMI as well as age and given a single capsule of either 0·47 g of Mirtoselect® (a standardised bilberry extract (36 % (w/w) anthocyanins)) which equates to about 50 g of fresh bilberries formulated in gelatin capsules or a control capsule consisting of microcrystalline cellulose in an opaque gelatin capsule, followed by oral glucose tolerance testing (OGTT). The reverse procedure was conducted following a 2-week washout period. The volunteers were asked to consume a low-phytochemical diet 3 d before taking the capsule and for the 24 h after taking the capsule on both occasions. In addition the volunteers were asked to record what they ate over the same period in a food diary to ensure that they adhered to the low-phytochemical diet. Subjects were reimbursed travelling expenses on completion of the study.
Period: Overall Study
Arm/Group | Single Control Capsule First Then Bilberry Capsule | Single Bilberry Capsule First Then Control Capsule
Started | 4 (In a cross-over design, volunteers (n=8) were randomised and double blinded into two groups (n=4)) | 4 (In a cross-over design, volunteers (n=8) were randomised and double blinded into two groups (n=4))
Completed | 4 (In a cross-over design, volunteers (n=8) were randomised and double blinded into two groups (n=4)) | 4 (In a cross-over design, volunteers (n=8) were randomised and double blinded into two groups (n=4))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bilberry Capsule First, Then Control Capsule; Control Capsule First, Then Bilberry Capsule: In a cross-over design, eight volunteers were randomised and double-blinded into two groups matched for BMI as well as age and given a single capsule of either 0·47 g of Mirtoselect® (a standardised bilberry extract (36 % (w/w) anthocyanins)) which equates to about 50 g of fresh bilberries formulated in gelatin capsules or a control capsule consisting of microcrystalline cellulose in an opaque gelatin capsule, followed by oral glucose tolerance testing (OGTT). The reverse procedure was conducted following a 2-week washout period. The volunteers were asked to consume a low-phytochemical diet 3 d before taking the capsule and for the 24 h after taking the capsule on both occasions. In addition the volunteers were asked to record what they ate over the same period in a food diary to ensure that they adhered to the low-phytochemical diet. Subjects were reimbursed travelling expenses on completion of the study.
- Total: Total of all reporting groups
Arm/Group | Bilberry Capsule First, Then Control Capsule | Control Capsule First, Then Bilberry Capsule | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (5) | 62 (5) | 62 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 4 | 8
BMI [Mean (Standard Deviation); unit: Kg/m2] | 30 (4) | 30 (4) | 30 (4)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose iAUC (Incremental Area Under the Curve; mM*Min)
Description: Volunteers were fasted (10-12 h) overnight before the OGTT. Venous blood samples were taken through an indwelling cannula inserted into a forearm vein at -15, -10 and -5 (fasted) and at 15, 30, 45, 60, 90, 120, 150 and 300 min after consuming 75 g of Polycal liquid (carbohydrate, 61·9%; polysaccharide, 49·2
  %; sugars, 12·2%; glucose, 0·6%; maltose, 11·6%; http://www. nutricia.co.uk). Polycal was selected as the main carbohydrate as it is in the form of polysaccharides and this is closer to normal dietary consumption than glucose only.The volunteers consumed the appropriate capsule (0 min), glucose load and a further sample of water (70 ml) within 3 min.
  For those volunteers taking the control capsule, additional sugar (fructose and dextrose/glucose) was added double-blinded to the water to match the free sugar content of the Mirtoselect® capsules. Movement during the 300 min OGTT was kept to a minimum.
Time Frame: Plasma was collected at -15, -10 and -5 (fasted) and at 15, 30, 45, 60, 90, 120, 150 and 300 min post capsule
Measure: Mean (Standard Error); unit: glucose iAUC (mM*min)
Groups:
- Single Placebo Capsule; Single Blaeberry Capsule: In a cross-over design, volunteers (n 8) were randomised and double-blinded into two groups matched for BMI as well as age and given a single capsule of either 0·47 g of Mirtoselect® (a standardised bilberry extract (36 % (w/w) anthocyanins)) which equates to about 50 g of fresh bilberries formulated in gelatin capsules or a control capsule consisting of microcrystalline cellulose in an opaque gelatin capsule, followed by oral glucose tolerance testing (OGTT). The reverse procedure was conducted following a 2-week washout period. The volunteers were asked to consume a low-phytochemical diet 3 d before taking the capsule and for the 24 h after taking the capsule on both occasions. In addition the volunteers were asked to record what they ate over the same period in a food diary to ensure that they adhered to the low-phytochemical diet. Subjects were reimbursed travelling expenses on completion of the study.
Arm/Group | Single Placebo Capsule | Single Blaeberry Capsule
Number analyzed (Participants) | 8 | 8
glucose iAUC (mM*min) | 836 (97) | 693 (103)
Statistical Analysis 1: Comparison: Single Placebo Capsule vs Single Blaeberry Capsule; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — For the incremental area under the curve (AUCi), only the extent of interpolated values above baseline contributed. Values obtained following the control and extract capsules were compared by paired t-tests

2. Primary Outcome: Plasma Insulin iAUC (Incremental Area Under the Curve; ng/ml*Min)
Description: Volunteers were fasted (10-12 h) overnight before the OGTT. Venous blood samples were taken through an indwelling cannula inserted into a forearm vein at -15, -10 and -5 (fasted) and at 15, 30, 45, 60, 90, 120, 150 and 300 min after consuming 75 g of Polycal liquid (carbohydrate, 61•9%; polysaccharide, 49•2
  %; sugars, 12•2%; glucose, 0•6%; maltose, 11•6%; http://www. nutricia.co.uk). Polycal was selected as the main carbohydrate as it is in the form of polysaccharides and this is closer to normal dietary consumption than glucose only.The volunteers consumed the appropriate capsule (0 min), glucose load and a further sample of water (70 ml) within 3 min.
  For those volunteers taking the control capsule, additional sugar (fructose and dextrose/glucose) was added double-blinded to the water to match the free sugar content of the Mirtoselect® capsules. Movement during the 300 min OGTT was kept to a minimum.
Time Frame: Plasma was collected at -15, -10 and -5 (fasted) and at 15, 30, 45, 60, 90, 120, 150 and 300 min after the capsule
Measure: Mean (Standard Error); unit: insulin iAUC (ng/ml*min)
Groups:
- Single Control Capsule; Single Bilberry Capsule: In a cross-over design, volunteers (n 8) were randomised and double-blinded into two groups matched for BMI as well as age and given a single capsule of either 0·47 g of Mirtoselect® (a standardised bilberry extract (36 % (w/w) anthocyanins)) which equates to about 50 g of fresh bilberries formulated in gelatin capsules or a control capsule consisting of microcrystalline cellulose in an opaque gelatin capsule, followed by oral glucose tolerance testing (OGTT). The reverse procedure was conducted following a 2-week washout period. The volunteers were asked to consume a low-phytochemical diet 3 d before taking the capsule and for the 24 h after taking the capsule on both occasions. In addition the volunteers were asked to record what they ate over the same period in a food diary to ensure that they adhered to the low-phytochemical diet. Subjects were reimbursed travelling expenses on completion of the study.
Arm/Group | Single Control Capsule | Single Bilberry Capsule
Number analyzed (Participants) | 8 | 8
insulin iAUC (ng/ml*min) | 358 (131) | 294 (113)
Statistical Analysis 1: Comparison: Single Control Capsule vs Single Bilberry Capsule; Test type: Superiority or Other; p = 0.028, t-test, 2 sided — For incremental area under the curve (AUCi), only the extent of interpolated values above baseline contributed. Values obtained following the control and extract capsules were compared by paired t-tests

3. Secondary Outcome: Bioavailability in Plasma
Description: To measure the amount of anthocyanins and phenolic-derived metabolites by liquid chromatography mass spectrometry (LC-MS) being absorbed from the gut and excreted following the single intervention.
Time Frame: Plasma will also be collected -15,-10, -5, 15, 30, 45, 60, 90, 120, 150, and 300 minutes and 24 hours post intervention
Reporting Status: Not Posted, anticipated posting 2022-09

4. Secondary Outcome: Bioavailability in Urine
Description: as for outcome 3
Time Frame: Urine will also be collected (if possible) 0, 1, 3 and 5 hours, with all urine collected within the 24 hour time period post intervention
Reporting Status: Not Posted, anticipated posting 2022-09

ADVERSE EVENTS:
Arm/Group | Single Bilberry Capsule | Single Placebo Capsule
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes